CLINICAL TRIAL: NCT02865369
Title: Regression of Liver Fibrosis Assessed by Transient Elastography After Daclatasvir and Asunaprevir Combined Treatment in Advanced Fibrotic/Cirrhotic Patients With Chronic Hepatitis C Genotype 1b Infection
Brief Title: Regression of Liver Fibrosis After Daclatasvir and Asunaprevir Treatment
Acronym: RELIF-C
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sang Gyune Kim (Other)
Collaborators: Seoul National University Boramae Hospital (Other); Severance Hospital (Other); Inha University Hospital (Other); Korea University (Other); Gachon University Gil Medical Center (Other); Hanyang University Seoul Hospital (Other); Ewha Womans University Mokdong Hospital (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Sang Gyune Kim, Professor, Soonchunhyang University Hospital
Organization: Soonchunhyang University Hospital (Other)
Other Study IDs: AI444-392
Record Dates: First submitted 2016-08-03; First posted 2016-08-12 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Chronic Hepatitis C
Keywords: chronic hepatitis C; Daclatasvir; Asunaprevir; fibrosis; transient elastography
MeSH Terms: conditions — Hepatitis C, Chronic; Fibrosis | interventions — daclatasvir; asunaprevir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — 8cc serum sample for the evaluation of direct liver fibrosis marker
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Daclatasvir plus Asunaprevir treatment: Among patients taking Daclatasvir and Asunaprevir combined treatment and having advanced liver fibrosis assessed by transient elastography
  Interventions: Drug: Daclatasvir and Asunaprevir

INTERVENTIONS:
Drug: Daclatasvir and Asunaprevir — Daclatasvir and Asunaprevir combined treatment will not be assigned to the enrolled patients, but the patients who are treated with Daclatasvir and Asunaprevir will be included in this observational study.
  Other Names: Daclatasvir and Asunaprevir combined treatment for 24 weeks

SUMMARY:
A study on regression of liver fibrosis assessed by transient elastography after Daclatasvir and Asunaprevir combined treatment in advanced fibrotic/cirrhotic patients with chronic hepatitis C genotype 1b Infection

DETAILED DESCRIPTION:
The measurement of liver stiffness by transient elastography (TE) has been shown to correlate with the hepatic fibrosis stage and to have considerable accuracy for the diagnosis of cirrhosis in patients with chronic hepatitis C. Previous studied reported that liver stiffness is significantly reduced in SVR patients with pegylated interferon (IFN) and ribavirin treatment. Once a patient achieve sustained virological response (SVR), and resultingly lower liver stiffness score than baseline value, it is believed that he will have a better long-term outcome due to the improvement of liver fibrosis.

Daclatasvir(DCV) and Asunaprevir(ASV) combined treatment showed a greater SVR rate in CHC compared to IFN based therapy. The investigators hypothesize that DCV and ASV combined treatment may achieve the improvement of liver stiffness measured by TE and a more favorable clinical outcomes in patients with advanced liver fibrosis. The investigators will also compare the change of fibrosis stage assessed by TE between this study subjects and those treated with other DAA agents during same observational period.

ELIGIBILITY:
Inclusion Criteria:

* Chronically infected with Hepatitis C virus genotype 1b
* HCV RNA ≥ 10^4 IU/mL (10,000 IU/mL)
* Chronic Hepatitis C with advanced fibrosis or cirrhosis (defined as ≥F3, ≥8 kilopascals)
* Treatment-naïve or those who previously failed to treatment with peg-interferon alfa and ribavirin
* Women of childbearing potential (WOCBP) and men, who use effective methods of birth control

Exclusion Criteria:

* Patients with baseline key NS5A RAVs (Y93 and/or L31)
* Estimated GFR < 30mL/min without hemodialysis
* Alanine aminotransferase (ALT) > 100 IU/L
* Coinfection with other hepatitis virus or human immunodeficiency virus
* A daily alcohol intake >30 g
* Decompensated liver disease or hepatocellular carcinoma, liver or any other organ transplantation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Genotype 1b, advanced fibrotic/cirrhotic Korean patients with chronic hepatitis C aged over 18, without baseline NS5A RAVs (Y93 and/or L31)
Sampling Method: Probability Sample
Enrollment: 103 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The change of liver fibrosis stage at 48 weeks assessed by transient elastography in patients treated with Daclatasvir and Asunaprevir | baseline to 48weeks
  To compare the change of liver fibrosis stage (defined as F3, ≥8; F4, ≥12) assessed by transient elastography between baseline and 48 weeks in advanced fibrotic/cirrhotic Chronic Hepatitis C patients who achieved sustained virological response with Daclatasvir and Asunaprevir combined treatment

SECONDARY OUTCOMES:
Proportion of patients who were treated with Daclatasvir and Asunaprevir achieved SVR12 assessed by HCV RNA | baseline to 36 weeks
Proportion of patients who maintained sustained virologic response at SVR24, SVR72, SVR120, SVR168, and SVR216. | baseline to 48weeks, 96weeks, 144weeks, 192weeks, 240weeks
The change of liver fibrosis stage assessed by transient elastography at 96weeks, 144weeks, 192weeks, 240weeks in patients treated with Daclatasvir and Asunaprevir | baseline to 96weeks, 144weeks, 192weeks, 240weeks
The change of AST to Platelet Ratio Index | baseline to 48weeks, 96weeks, 144weeks, 192weeks, 240weeks
  APRI = [(AST/upper limit of normal)/platelet count]x100
The change of Fibrosis 4 (Fib-4) index | baseline to 48weeks, 96weeks, 144weeks, 192weeks, 240weeks
  FIB-4 = age (years) × AST [IU/L] / [platelet count × sqr(ALT [IU/L])]
Comparison of change of liver fibrosis stage assessed by transient elastography between Daclatasvir and Asunaprevir combined treatment versus other DAA treatment | baseline to 48weeks, 96weeks, 144weeks, 192weeks, 240weeks
  Comparison of change of liver fibrosis stage assessed by transient elastography at 48weeks, 96weeks, 144weeks, 192weeks, 240weeks between Daclatasvir and Asunaprevir combined treatment versus other DAA treatment during same observational period
Comparison of the incidence of hepatocellular carcinoma or liver cirrhosis complications between Daclatasvir and Asunaprevir combined treatment versus other DAA treatment | baseline to 48weeks, 96weeks, 144weeks, 192weeks, 240weeks
  Compare the incidence of hepatocellular carcinoma or liver cirrhosis complications at 48weeks, 96weeks, 144weeks, 192weeks, 240weeks between Daclatasvir and Asunaprevir combined treatment versus other Direct antiviral agents during same observational period
The change of Fibrometer score | baseline to 48weeks, 96weeks, 144weeks, 192weeks, 240weeks
  alpha2 macroglobulin, GGT, AST, ALT, prothrombin index, urea, platelet count

CONTACTS AND LOCATIONS:
Overall Officials: Sang Gyune Kim, Professor, Principal Investigator — Soonchunhyang University Hospital
Locations (10):
- South Korea (10):
  - Soonchunhyang University Cheonan Hospital, Cheonan, Chungcheongnam-do
  - Korea University Ansan Hospital, Ansan, Gyeonggi-do
  - Soon Chun Hyang University Bucheon Hospital, Bucheon-si, Gyeonggi-do
  - Inha University Hospital, Jung-gu, Incheon
  - Gachon University Gil Medical Center, Incheon
  - Severance hospital, Seoul
  - Soonchunhyang University Hospital, Seoul
  - Hanyang university hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Wonju severance christian hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ziol M, Handra-Luca A, Kettaneh A, Christidis C, Mal F, Kazemi F, de Ledinghen V, Marcellin P, Dhumeaux D, Trinchet JC, Beaugrand M. Noninvasive assessment of liver fibrosis by measurement of stiffness in patients with chronic hepatitis C. Hepatology. 2005 Jan;41(1):48-54. doi: 10.1002/hep.20506. PMID 15690481
- [Background] Hezode C, Castera L, Roudot-Thoraval F, Bouvier-Alias M, Rosa I, Roulot D, Leroy V, Mallat A, Pawlotsky JM. Liver stiffness diminishes with antiviral response in chronic hepatitis C. Aliment Pharmacol Ther. 2011 Sep;34(6):656-63. doi: 10.1111/j.1365-2036.2011.04765.x. Epub 2011 Jul 13. PMID 21752038
- [Background] Arima Y, Kawabe N, Hashimoto S, Harata M, Nitta Y, Murao M, Nakano T, Shimazaki H, Kobayashi K, Ichino N, Osakabe K, Nishikawa T, Okumura A, Ishikawa T, Yoshioka K. Reduction of liver stiffness by interferon treatment in the patients with chronic hepatitis C. Hepatol Res. 2010 Apr;40(4):383-92. doi: 10.1111/j.1872-034X.2009.00618.x. Epub 2010 Mar 4. PMID 20236358
- [Background] Wang JH, Changchien CS, Hung CH, Tung WC, Kee KM, Chen CH, Hu TH, Lee CM, Lu SN. Liver stiffness decrease after effective antiviral therapy in patients with chronic hepatitis C: Longitudinal study using FibroScan. J Gastroenterol Hepatol. 2010 May;25(5):964-9. doi: 10.1111/j.1440-1746.2009.06194.x. PMID 20546451
- [Background] Crisan D, Radu C, Grigorescu MD, Lupsor M, Feier D, Grigorescu M. Prospective non-invasive follow-up of liver fibrosis in patients with chronic hepatitis C. J Gastrointestin Liver Dis. 2012 Dec;21(4):375-82. PMID 23256120
- [Background] Bourliere, Marc, et al.
- [Derived] Yoo HW, Park JY, Kim SG, Jung YK, Lee SH, Kim MY, Jun DW, Jang JY, Lee JW, Kwon OS. Regression of liver fibrosis and hepatocellular carcinoma development after HCV eradication with oral antiviral agents. Sci Rep. 2022 Jan 7;12(1):193. doi: 10.1038/s41598-021-03272-1. PMID 34996920